CLINICAL TRIAL: NCT02946086
Title: Effect of Rehabilitation in Deficiencies, Activities Limitations and Restrictions of the Participation of the Children Presenting Neurological Lesions. Impact of Contextual Factors on the Functioning of These Patients. Part II
Brief Title: Effect of HABIT-ILE on Visuo-spatial Attention of Children With Unilateral CP
Acronym: HABIT-ILE_CP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Yannick Bleyenheuft, Professor, Université Catholique de Louvain
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B403201316810
Record Dates: First submitted 2015-12-21; First posted 2016-10-26 (Estimated); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Cerebral Palsy
Keywords: motor skill learning, visuo-spatial attention
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- prismatic adaptation (Experimental): Including 8 hours of therapy with prismatic adaptation wearing prismatic goggles during bimanual intensive and locomotor intensive intervention (HABIT-ILE).
  Interventions: Behavioral: HABIT-ILE with prismatic adaptation
- sham goggles (Active Comparator): Including 8 hours of therapy wearing "sham goggles" during bimanual intensive and locomotor intensive intervention (HABIT-ILE).
  Interventions: Behavioral: HABIT-ILE without prismatic adaptation

INTERVENTIONS:
Behavioral: HABIT-ILE with prismatic adaptation — Bimanual and locomotor intensive intervention for 90h including 8 hours of prismatic adaptation
  Arms: prismatic adaptation
Behavioral: HABIT-ILE without prismatic adaptation — Bimanual and locomotor intensive intervention for 90h including 8 hours of prismatic adaptation wearing sham goggles.
  Arms: sham goggles

SUMMARY:
This study aims to investigate the changes induced by HABIT-ILE in impairments, activity and participation of children with unilateral CP, as well as neuroplastic changes induced by the treatment. Visuospatial deficits will be investigated and the effect of prismatic adaptation will be measured.

DETAILED DESCRIPTION:
This study aims to investigate the changes induced by HABIT-ILE at the 3 levels of the international classification of functioning and health (ICF) in children with unilateral CP, as well as neuroplastic changes induced by the treatment. Visuospatial deficits will be investigated and the effect of prismatic adaptation will be measured.

ELIGIBILITY:
Inclusion Criteria:

* unilateral CP
* minimal ability to pick an light object from a table
* age 5-18

Exclusion Criteria:

* no active seizure
* no botox or orthopedic intervention in the 6 months preceding the study or during the study

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2013-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
changes in star cancellation | at baseline and after 90 hours/two weeks of intensive bimanual intervention
  number of little stars omitted in a frame including many stars of different size
change in "Ogden Figure" test | at baseline and after 90 hours/two weeks of intensive bimanual intervention
  number of elements omitted when reproducing a drawing
changes in line bissection | at baseline and after 90 hours/two weeks of intensive bimanual intervention
  deviation from midline during line section
visuo-spatial pointing | at baseline and after 90 hours/two weeks of intensive bimanual intervention
  pointing in a blind box in the direction of a visual cue, measuring the deviation from midline
proprioceptive pointing | at baseline and after 90 hours/two weeks of intensive bimanual intervention
  pointing without any visual feedback in the direction of body midline and measuring deviation

SECONDARY OUTCOMES:
Jebsen-Taylor test of hand function | at baseline and after 90 hours/two weeks of intensive bimanual intervention
  Manual dexterity measured with objects of everyday life, measure=time to manipulate objects
functional magnetic resonance imaging (fMRI) | at baseline and after 90 hours/two weeks of intensive bimanual intervention
  cortical activation (changes in voxels activation)
Box and blocks | at baseline and after 90 hours/two weeks of intensive bimanual intervention
  number of blocks manipulated in one minute
Assisting Hand Assessment | at baseline and after 90 hours/two weeks of intensive bimanual intervention
  help provided by the paretic hand to the non-paretic one in bimanual coordination
"ABILHAND-Kids" questionnaire | at baseline and after 90 hours/two weeks of intensive bimanual intervention
  parents-reported questionnaire measuring manual ability
"ACTIVLIM-CP" questionnaire | at baseline and after 90 hours/two weeks of intensive bimanual intervention
  parents-reported questionnaire measuring global activity performance
Canadian Occupationnal Performance Measure | at baseline and after 90 hours/two weeks of intensive bimanual intervention
  setting therapeutic goals with parents and measuring both performance and satisfaction (%)
diffusion tensor imaging (DDTI) | at baseline and after 90 hours/two weeks of intensive bimanual intervention
  measuring changes in white matter tracts (fractional anisotropy, number of voxels)

CONTACTS AND LOCATIONS:
Overall Officials: Yannick Bleyenheuft, PhD, Principal Investigator — Institute of Neuroscience, Université catholique de Louvain
Locations (1):
- Bleyenheuft Yannick, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No